CLINICAL TRIAL: NCT03972735
Title: Randomized Controlled Study on the Efficacy of the NECT Program (Cognitive Therapy and Narrative Development) on Improving Social Functioning in People With Severe Psychic Disorders
Brief Title: Assessment of the Effectiveness of the NECT Program
Acronym: NECT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Center Alpes-Isère (Other)
Collaborators: Hôpital le Vinatier (Other); University Hospital, Grenoble (Other); Clinique du Dauphiné (Unknown); CH Annecy Genevois (Other); University Hospital, Clermont-Ferrand (Other); Centre Hospitalier Esquirol (Other); Centre Hospitalier Universitaire de Nice (Other); CHS LE VALMONT (Unknown); University Hospital, Caen (Other); University Hospital, Geneva (Other); University Hospital, Montpellier (Other)
Responsible Party: Principal Investigator, Dr Julien Dubreucq, Medical doctor, Hospital Center Alpes-Isère
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2018-A03237-48
Record Dates: First submitted 2019-05-31; First posted 2019-06-04 (Actual); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: Schizophrenia; Bipolar Disorder; Borderline Personality Disorder; Social Function; Self-stigma
MeSH Terms: conditions — Schizophrenia; Bipolar Disorder; Borderline Personality Disorder; Social Adjustment | interventions — Neuropsychological Tests

STUDY DESIGN:
Intervention Model Description: stepped-wedge
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NECT + follow up (Experimental): Narrative Development and Cognitive Therapy (NECT) is a 12 session group-based manualized intervention combining psychoeducation, cognitive restructuring and narrative enhancement. The 2 hours sessions are conducted by two trained facilitators.
  Interventions: Other: Psychiatric interview; Other: Clinical, diagnostic and functional evaluation; Other: neuropsychological assessment; Other: NECT PROGRAM
- TAU (Placebo Comparator): * Drug treatment (antipsychotic, mood stabilizing) for people with schizophrenia or with bipolar disorder
  * Support in day-care hospital
  * No intervention specifically targeting self-stigma reduction or improvements in social functioning (social cognitive remediation or social skills training)
  Interventions: Other: Psychiatric interview; Other: Clinical, diagnostic and functional evaluation; Other: neuropsychological assessment; Other: NECT PROGRAM

INTERVENTIONS:
Other: Psychiatric interview — PANSS, MADRS, PSP, YMRS
Other: Clinical, diagnostic and functional evaluation — ISMI, STORI, SERS, S-QOL, WEWMBS, BIRCHWOOD, MARS
Other: neuropsychological assessment — WAIS IV, BEM 144, TMT A, TMT B, D2-R, V-LIS
Other: NECT PROGRAM — Narrative Development and Cognitive Therapy (NECT) is a 12 session group-based manualized intervention combining psychoeducation, cognitive restructuring and narrative enhancement. The 2h sessions are conducted by two trained facilitators.

SUMMARY:
Self-stigma refers to the transformation process wherein a person's previously held social identity is progressively replaced by a devalued and stigmatized view of oneself termed "illness identity". Self-Stigma is a severe problem in Serious Mental Illness (SMI). Self-stigma prevalence is high (41.7% of the 1229 participants with SZ and 21.7% of the 1182 participants with mood disorders had moderate to high levels of IS in the GAMIAN-Europe study). Self-stigma was negatively associated with self-esteem, social function, wellbeing, quality of life or personal recovery and positively associated with psychiatric symptoms and depression. Several psychosocial interventions (mostly combinations of psychoeducation and cognitive behaviour therapy) have been designed to reduce self-stigma and its impact on clinical and functional outcomes, with preliminary effects on self-stigma, insight and self-efficacy.

Narrative Enhancement and Cognitive Therapy (NECT) is a manualized structured 20-session group-based intervention . Conducted by two trained facilitators the sessions combine psychoeducation, cognitive restructuring and story-telling exercises to reduce self-stigma. Developed in USA, NECT was adapted in Israel and Sweden. NECT showed effectiveness in reducing self-stigma and in improving self-esteem and quality of life. Despite being effective on changing coping strategies, NECT effectiveness on social function is still unclear.

The present study aims to validate NECT French adaptation and to evaluate its effectiveness on social function, self-stigma, psychiatric symptoms, self-esteem, wellbeing, quality of life and personal recovery in SMI participants (schizophrenia, bipolar disorder, borderline personality disorder)

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia, schizoaffective disorder, schizotypal disorder, schizophreniform disorder, bipolar I or II disorder, borderline personality disorder (DSM-V criteria, APA, 2013).
* Clinical stability since 3 months (total PANSS score <120, MADRS score <15 and YMRS <12 for patients with schizophrenia and MADRS score <15 and YMRS <12 for patients with bipolar disorder).
* Patients who gave informed consent to participate in the study.
* Affiliated to a social security scheme or beneficiary of such a scheme.

Exclusion Criteria:

* Pregnant or lactating women.
* Criteria relating to the associated pathologies entailing particular risks:
* Neurological disorders of vascular, infectious or neurodegenerative origin.
* Taking somatic drugs with a cerebral or mental impact (eg corticosteroids).
* Presence of an associated intellectual disability.
* Prohibited treatments and procedures:
* Subject in exclusion period of another study.
* Simultaneous participation in other programs having an impact on social functioning or self-stigmatization: remediation of social cognition, individual and group care targeting self-stigmatization and training in social skills.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-02-10 (Actual); Primary Completion 2022-09-01 (Estimated); Study Completion 2023-04-01 (Estimated)

PRIMARY OUTCOMES:
Personal and Social Performance Scale | Changes between baseline function, at 6, 12 and 18 months of follow-up
  Changes in the aggregates (average) of standardized performance levels : z-scores of social function (0 to 100) after NECT Program

SECONDARY OUTCOMES:
Internalized Stigma of Mental Illness (ISMI) scale | Changes between baseline function, at 6, 12 and 18 months of follow-up
  self-assessment of internalized stigma (mean score of total self-stigma ranging from 1 to 4)
Positive and Negative Symptoms Scale for Schizophrenia (PANSS) | Changes between baseline function, at 6, 12 and 18 months of follow-up
  Changes in the aggregates (average) of standardized performance levels : z-scores of positive and negative symptoms (minimum score 30- maximum score 210) of schizophrenia after NECT Program
MADRS (Montgomery-Asberg Depression Rating) | Changes between baseline function, at 6, 12 and 18 months of follow-up
  Changes in the aggregates (average) of standardized performance levels
BIRCHWOOD INSIGHT SCALE | Changes between baseline function, at 6, 12 and 18 months of follow-up
  Changes in the aggregates (average) of standardized performance levels
MARS (Medication Adherence Rating Scale) | Changes between baseline function, at 6, 12 and 18 months of follow-up
  self-assesment of adherence into treatment (minimum 1-maximum 10)
WEMWBS (Warwick Edinburgh Mental Well Being Scale) ) | Changes between baseline function, at 6, 12 and 18 months of follow-up
  self assessment of mental well being
SERS (Self-Esteem Rating Scale) | Changes between baseline function, at 6, 12 and 18 months of follow-up
  Changes in the aggregates (average) of standardized performance levels : z-scores (minimum score 10-maximum score 70) in self-assessment of self-esteem
S-QOL (Subjective Quality of Life) | Changes between baseline function, at 6, 12 and 18 months of follow-up
  sel-assessment of quality of life (minimum 0, maximum 100)
STORI Stages of Recovery Instrument | Changes between baseline function, at 6, 12 and 18 months of follow-up
  Self-assessment of personal recovery (maximum stage of recovery ranging from 0 to 5

CONTACTS AND LOCATIONS:
Overall Officials: Julien JD DUBREUCQ, MD, Principal Investigator — Hospital Center Alpes-Isère
Locations (11):
- France (10):
  - Ch Annecy-Genevois, Annecy, AURA
  - Ch Le Vinatier, Bron, Aura
  - CHU de CLERMONT-FERRAND, Clermont-Ferrand, AURA
  - University Hospital, Grenoble, Grenoble, AURA
  - CHS Esquirol, Limoges, Aura
  - Clinique du Dauphiné, Seyssins, AURA
  - Chs Le Valmont, Valence, AURA
  - E.P.S.M. Ariane, Caen, Normandy
  - Hopital La Colombière, University Hospital Montpellier, Montpellier, Occitanie
  - Hospital Center SAINTE MARIE, Nice, Paca
- Service des Specialités psychiatriques, Geneva, Switzerland

REFERENCES:
- [Background] Bellack AS, Brown SA. Psychosocial treatments for schizophrenia. Curr Psychiatry Rep. 2001 Oct;3(5):407-12. doi: 10.1007/s11920-996-0035-x. PMID 11559478
- [Background] Brohan E, Elgie R, Sartorius N, Thornicroft G; GAMIAN-Europe Study Group. Self-stigma, empowerment and perceived discrimination among people with schizophrenia in 14 European countries: the GAMIAN-Europe study. Schizophr Res. 2010 Sep;122(1-3):232-8. doi: 10.1016/j.schres.2010.02.1065. Epub 2010 Mar 26. PMID 20347271
- [Background] Corrigan PW, Larson JE, Rusch N. Self-stigma and the "why try" effect: impact on life goals and evidence-based practices. World Psychiatry. 2009 Jun;8(2):75-81. doi: 10.1002/j.2051-5545.2009.tb00218.x. PMID 19516923
- [Background] Corrigan PW, Kosyluk KA, Rusch N. Reducing self-stigma by coming out proud. Am J Public Health. 2013 May;103(5):794-800. doi: 10.2105/AJPH.2012.301037. Epub 2013 Mar 14. PMID 23488488
- [Background] Dixon LB, Dickerson F, Bellack AS, Bennett M, Dickinson D, Goldberg RW, Lehman A, Tenhula WN, Calmes C, Pasillas RM, Peer J, Kreyenbuhl J; Schizophrenia Patient Outcomes Research Team (PORT). The 2009 schizophrenia PORT psychosocial treatment recommendations and summary statements. Schizophr Bull. 2010 Jan;36(1):48-70. doi: 10.1093/schbul/sbp115. Epub 2009 Dec 2. PMID 19955389
- [Background] Fung KM, Tsang HW, Cheung WM. Randomized controlled trial of the self-stigma reduction program among individuals with schizophrenia. Psychiatry Res. 2011 Sep 30;189(2):208-14. doi: 10.1016/j.psychres.2011.02.013. Epub 2011 Mar 5. PMID 21377738
- [Background] Lysaker PH, Bond G, Davis LW, Bryson GJ, Bell MD. Enhanced cognitive-behavioral therapy for vocational rehabilitation in schizophrenia: Effects on hope and work. J Rehabil Res Dev. 2005 Sep-Oct;42(5):673-82. doi: 10.1682/jrrd.2004.12.0157. PMID 16586193
- [Background] Lysaker PH, Roe D, Yanos PT. Toward understanding the insight paradox: internalized stigma moderates the association between insight and social functioning, hope, and self-esteem among people with schizophrenia spectrum disorders. Schizophr Bull. 2007 Jan;33(1):192-9. doi: 10.1093/schbul/sbl016. Epub 2006 Aug 7. PMID 16894025
- [Background] Rusch N, Lieb K, Bohus M, Corrigan PW. Self-stigma, empowerment, and perceived legitimacy of discrimination among women with mental illness. Psychiatr Serv. 2006 Mar;57(3):399-402. doi: 10.1176/appi.ps.57.3.399. PMID 16525000
- [Background] Vauth R, Kleim B, Wirtz M, Corrigan PW. Self-efficacy and empowerment as outcomes of self-stigmatizing and coping in schizophrenia. Psychiatry Res. 2007 Feb 28;150(1):71-80. doi: 10.1016/j.psychres.2006.07.005. Epub 2007 Jan 30. PMID 17270279
- [Background] Yanos PT, Roe D, Markus K, Lysaker PH. Pathways between internalized stigma and outcomes related to recovery in schizophrenia spectrum disorders. Psychiatr Serv. 2008 Dec;59(12):1437-42. doi: 10.1176/ps.2008.59.12.1437. PMID 19033171
- [Result] Livingston JD, Boyd JE. Correlates and consequences of internalized stigma for people living with mental illness: a systematic review and meta-analysis. Soc Sci Med. 2010 Dec;71(12):2150-61. doi: 10.1016/j.socscimed.2010.09.030. Epub 2010 Oct 12. PMID 21051128
- [Result] Lucksted A, Drapalski AL, Brown CH, Wilson C, Charlotte M, Mullane A, Fang LJ. Outcomes of a Psychoeducational Intervention to Reduce Internalized Stigma Among Psychosocial Rehabilitation Clients. Psychiatr Serv. 2017 Apr 1;68(4):360-367. doi: 10.1176/appi.ps.201600037. Epub 2016 Dec 1. PMID 27903136
- [Result] Roe D, Hasson-Ohayon I, Mashiach-Eizenberg M, Derhy O, Lysaker PH, Yanos PT. Narrative enhancement and cognitive therapy (NECT) effectiveness: a quasi-experimental study. J Clin Psychol. 2014 Apr;70(4):303-12. doi: 10.1002/jclp.22050. Epub 2013 Oct 2. PMID 24114797
- [Derived] Dubreucq J, Faraldo M, Abbes M, Ycart B, Richard-Lepouriel H, Favre S, Jermann F, Attal J, Bakri M, Cohen T, Cervello C, Chereau I, Cognard C, De Clercq M, Douasbin A, Giordana JY, Giraud-Baro E, Guillard-Bouhet N, Legros-Lafarge E, Polosan M, Pouchon A, Rolland M, Rainteau N, Roussel C, Wangermez C, Yanos PT, Lysaker PH, Franck N. Narrative enhancement and cognitive therapy (NECT) to improve social functioning in people with serious mental illness: study protocol for a stepped-wedge cluster randomized controlled trial. Trials. 2021 Feb 8;22(1):124. doi: 10.1186/s13063-021-05067-1. PMID 33557924